CLINICAL TRIAL: NCT04032782
Title: A First-in-Human, Double-blind, Randomized, Placebo-controlled, Single Ascending Dose Study to Assess Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of HM15136(Efpegerglucagon) in Healthy Subjects
Brief Title: A First-in-Human, Study to Assess Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of HM15136(Efpegerglucagon) in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM-GCG-101
Record Dates: First submitted 2018-11-16; First posted 2019-07-25 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Pharmacology
MeSH Terms: interventions — HM15136

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HM15136 (Experimental)
  Interventions: Drug: HM15136
- Placebo of HM15136 (Placebo Comparator)
  Interventions: Drug: Placebo of HM15136

INTERVENTIONS:
Drug: HM15136 — 10 mg/mL as protein in prefilled syringes
  Arms: HM15136
Drug: Placebo of HM15136 — Placebo in prefilled syringes
  Arms: Placebo of HM15136

SUMMARY:
This is a double-blind, randomized, placebo controlled, single ascending dose (SAD) study to investigate the safety, tolerability, PK and PD of the SC administration of HM15136 in healthy subjects.

The study will be conducted in approximately 5 sequential dosing cohorts, enrolling 8 subjects per cohort. Subjects will be randomized to HM15136 or placebo in a ratio of 6:2 (6 active, 2 placebo).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index ≥ 18.5 and ≤ 27 kg/m2 and with a weight ≥ 50 kg

Exclusion Criteria:

* with personal or family history of hypercoagulability or thromboembolic disease
* has had treatment with any incretin therapy
* has FPG < 70 or > 110 mg/dL

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

PRIMARY OUTCOMES:
Adverse Event | Day 30
  Incidence of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea